CLINICAL TRIAL: NCT06809725
Title: Validation of the SPARK Scan Cognitive Status Indicator Software Concordance With Clinical Diagnosis in Humans With Unimpaired, Mild Cognitive Impairment and Dementia Status, With and Without Alzheimer's Disease
Brief Title: Software Validation Study-Cognitive Status Indicator
Acronym: REMIND-V
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Neuro Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1002; 2R44AG078039-02 (NIH)
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Dementia
Keywords: Alzheimer; dementia; Mild Cognitive Impairment; EEG
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: Software validation study (EEG used as data collection intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Dementia subjects (Experimental): EEG data from subjects are used to validate algorithm
  Interventions: Diagnostic Test: SPARK Cognitive Status Indicator (software support data collected via EEG)

INTERVENTIONS:
Diagnostic Test: SPARK Cognitive Status Indicator (software support data collected via EEG) — The SPARK Cognitive Status Indicator software (collected via EEG) is being validated to aid in the diagnosis of Alzheimer's disease in persons aged 65-90 with suspected cognitive impairment. The device, once validated, shall provide a clinician with a "positive" or "negative" output to indicate whether the subject's electroencephalogram (EEG) is consistent with EEGs of subjects diagnosed with Alzheimer's disease.

SUMMARY:
The SPARK Cognitive Status Indicator software uses an algorithm to assess a resting state EEG recording as being consistent with a cognitive status of unimpaired, mild cognitive impairment (MCI; MCI AD- or MCI AD+), or dementia (dementia AD-, or dementia AD+). This study will compare SPARK Cognitive Status Indicator output to Adjudication Committee panel-based diagnosis of cognitive status and Alzheimer's disease.

DETAILED DESCRIPTION:
Up to 600 subjects (and informants) may be enrolled and have a brain scan, cognitive, and blood assessments collected:

Visit 1-Screening:

-Salzburg (SDTP)- remote via telephone or video visit

Visit 2/3-Evaluations:

* EEG Scan (brain scan)
* Mini-Mental State Exam (MMSE)-at home visit
* Functional Assessment Staging Tool (FAST)- at home via video visit
* blood- Amyloid Beta 42/40 ratio, p tau- at laboratory or home visit There are three instances of subject engagement with the study team after informed consent. One, during screening which may be a remote visit and and two different home or remote visits (or laboratory visit). The study participation ends when all of the assessments have been collected. The total duration of subject participation should be no more than 2-3 days within a 90 day period.

The output of the investigational software used in the analysis to determine a identification of cognitive and Alzheimer's status based the data from the EEG scan shall be compared to the identification of cognitive and Alzheimer's status from a group of dementia specialists forming an Adjudication Committee which shall review all data (except for investigational device output).

ELIGIBILITY:
Inclusion Criteria:

Unimpaired subjects:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 65 to 90 at the time of consent
4. Have a Salzburg Dementia Test Prediction (SDTP) score >= 24.
5. Informant, available and willing (remotely or in-person) to provide information about subject cognitive functioning
6. No Medical History of cognitive impairment

Mild Cognitive Impairment subjects:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. 1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 65 to 90 at the time of consent
4. Have a Salzburg Dementia Test Prediction (SDTP) score < 24.
5. Informant, available and willing (remotely or in-person) to provide information about subject cognitive functioning
6. Suspected or diagnosed with a mild cognitive issue

Dementia subjects:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form-legally authorized representative or individual
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 65 to 90 at the time of consent
4. Have a Salzburg Dementia Test Prediction (SDTP) score < 24.
5. Informant, available and willing (remotely or in-person) to provide information about subject cognitive functioning
6. Exhibiting and diagnosed with moderate or severe cognitive issue

Informants:

To be eligible to participate as an informant in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form 2. Typically spends 2 or more hours per month with subject. 3. Available and willing (remotely or in-person) to provide information about subject cognitive functioning

-

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Currently experiencing a skin disease on scalp that would affect electrode contacts in the opinion of the user

-

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of SPARK Cognitive Status Indicator compared to Adjudicated cognitive status | Day 1
  Software output of investigational device shall be compared to the cognitive status as determined by an Adjudication Committee
Sensitivity of SPARK Cognitive Status Indicator when identifying Alzheimer's disease in impaired subjects | Day 1
  Software output sensitivity will be computed from device AD+ output compared to the Adjudication Committee findings of AD positive cases (MCI and dementia subjects)
Specificity of SPARK Cognitive Status Indicator when identifying Alzheimer's disease in impaired subjects | Day 1
  Software output specificity will be computed from device AD- output compared to the Adjudication Committee findings of AD negative cases (MCI and dementia subjects)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Yoder, PI, PhD, Principal Investigator — SPARK Neuro
Locations (1):
- Remote, Miami, Florida, United States